CLINICAL TRIAL: NCT02591069
Title: Vagus Nerve Stimulation in Patients With Chronic Consciousness Disorders
Brief Title: Vagal Nerve Stimulation in Coma Patients
Acronym: SNV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-833; 2014-A00125-42 (Other: ID-RCB)
Record Dates: First submitted 2015-10-06; First posted 2015-10-29 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Chronic Consciousness Disorders; Vegetative State; Minimally Conscious State; Akinetic Mutism
Keywords: Vagus nerve stimulation; vegetative state; minimally conscious state; akinetic mutism; consciousness; connectivity
MeSH Terms: conditions — Persistent Vegetative State; Akinetic Mutism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients will undergo the same procedure (Experimental)
  Interventions: Device: stimulation device

INTERVENTIONS:
Device: stimulation device — All patients included in the study will undergo baseline assessment of all measures before surgery (implantation of a vagus nerve stimulation device). A second baseline assessment will take place after surgery, before the beginning of the stimulation. Stimulation intensity will start at 0.25mA and increase progressively by 0.25mA each week until reaching 1mA. Then, intensity will be set at 1.5mA (recommended by manufacturer) and will stay to this level until the end of the trial. Experimenters will keep the right to modify these parameters depending on patients' reaction to the treatment.

SUMMARY:
Minimally Conscious (MCS) or Vegetative State (VS) are disorders of consciousness which often occur following traumatic brain injury or ischemia. These alterations result most of the time in patients' loss of autonomy and require long years of special care. No efficient therapy to improve patients' consciousness has been found so far. Investigators propose to use vagal nerve stimulation (VNS) to restore cortical activity and patients' embodied self. The investigators' main hypothesis is that VNS will reestablish the thalamo-cortical connectivity leading to an improvement of the consciousness state. To test this hypothesis, investigators will use behavioral measures as well as fMRI, PET scan and EEG to assess brain activity. Patients will be evaluated before and during eight months following implantation of the stimulation device.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years old
* Patients with history of cranial trauma, cerebrovascular accident, or other event leading to cerebral anoxia, suffering of chronic alteration of consciousness (Vegetative State, Minimally Conscious State, akinetic mutism). The diagnostic will be based on clinical scales
* Patients already having a neurophysiologic checkup (EEG)
* Patients breathing without invasive help, and who are in a stable medical state
* Patients with a history of disease of at least 6 months
* Patients without clinical evolution for several months
* Patients with social security
* Patients for whom a family member have signed a written consent

Exclusion Criteria:

* Patients with tracheotomy
* Pregnant women
* Intubated patients
* Patients with damaged vagus nerves
* Patients with pre existing neurological conditions other than the one responsible for the consciousness disorder
* Patients with medical complications
* Patients suffering of septic infection
* Patients with a significant dysphagia
* Patients with dyspnea or shortness of breath
* Patients with obstructive sleep apnea
* Patients with any conditions non authorized by the stimulating device manufacturer (Cyberonics)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change over time of clinical scores on the Coma Recovery Scale - Revised | First assessment one week before implantation second assessment 3 weeks after implantation, then once per week for a month starting one week after the beginning of stimulation; then once a month for 6 months.
  The primary outcome will be the change over time of patients' clinical state. Investigators will employ a widely used scale: Coma Recovery Scale - Revised. Patients will be evaluated by the same trained doctor. Results will be analyzed using a within subject design, each patients will be his own control. Investigators predict a progressive improvement after the onset of treatment, compared to the two pre-stimulation evaluations.

SECONDARY OUTCOMES:
Evaluation of brain activity changes using EEG | First assessment one week before implantation second assessment 3 weeks after implantation, then once per week for a month starting one week after the beginning of stimulation, then once a month for 6 months.
  EEG will allow investigators to monitor brain activity at rest as well as in response to various sensory stimuli. Investigators will measure changes in evoked potentials, source of activity and frequency power known to be altered in coma patients. In addition EEG will offer the opportunity to record brain activity while the stimulating device is on.
MRI (anisotropy and fibers density) evaluation of anatomo-connectivity changes | First assessment one week before implantation second assessment 3 weeks after implantation and then one, three and six months after the onset of stimulation.
  Investigators will use Diffusion Tensor Imaging (DTI) before and after VNS to evaluate anisotropy and anatomical connectivity between brain stem, thalamus and various cortical areas, especially regarding the thalamo-cortical loops. During the MRI exams the stimulation device will be turned off for safety reasons.
fMRI evaluation of bold signal resting state activity and functional connectivity changes | Firsts First assessment one week before implantation second assessment 3 weeks after implantation,, and then one, three and six months after the onset of stimulation.
  WInvestigators will perform resting state analysis of bold signal and functional connectivity to quantify reactivation of brain region after VNS and inter region communication, especially regarding the thalamo-cortical loops. During the fMRI exams the stimulation device will be turned off for safety reasons.
PET scan evaluation of brain metabolism (Glucose consumption) changes | One baseline assessment one week before stimulation and a second one after 3 months of stimulation.
  Investigators will use the radioligand Fluorodesoxyglucose [18F-FDG] to assess brain consumption of glucose. This measure is complementary to the one provided by fMRI and has already been used in coma patients. Moreover, thanks to a hybrid MRI/PET scanner, investigators will perform the two exams simultaneously to correlate these two measures in real time.
Monitoring heart rate variability | First assessment one week before implantation second assessment 3 weeks after implantation, then once per week for a month starting one week after the beginning of stimulation, then once a month for 6 months.
  Investigators hypothesize that VNS will modulate several physiological parameters, among those Heart Rate Variability, a marker of the balance between sympathetic and parasympathetic activity. Investigators will measure changes of high frequencies / low frequencies ratio.
: Monitoring changes of serum free serotonin concentration | First assessment one week before implantation second assessment 3 weeks after implantation, then once per week for a month starting one week after the beginning of stimulation, then once a month for 6 months.
  Vagus nerve is known to stimulate raphe nuclei, the region of serotonin synthesis. Investigators hypothesize that VNS will increase serum free serotonin concentration. Investigators will measure it using high performance liquid chromatography, and report the changes of values of serotonin concentration.
Monitoring changes of thermal reaction to emotional stimuli | First assessment one week before implantation second assessment 3 weeks after implantation, then once per week for a month starting one week after the beginning of stimulation, then once a month for 6 months.
  Investigators will use regulation of facial temperature as an index of consciousness. When humans react to emotions, the temperature of their face changes. This regulation is dependent on consciousness state, and therefore should vary across time in this protocol. Investigators will measure changes in temperature (°Celsius) of patients' face throughout the task.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Luauté, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Neurologique de Lyon Pierre Wertheimer, Bron, France